CLINICAL TRIAL: NCT04431492
Title: Effect of Anaesthesia and Surgery on Plasma Levels of Nitric Oxide and Basic Aminoacids
Brief Title: Effect of Anaesthesia on Basic Aminoacids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: 13700418
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Effect of Anaesthesia on Basic Aminoacids

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coronary artery bypass
  Interventions: Procedure: CABG
- thoracic surgery

INTERVENTIONS:
Procedure: CABG — aminoacids and NO levels
  Groups: coronary artery bypass

SUMMARY:
Basic amino acids are acids that contains amino groups more than carboxylic groups. At least five basic amino acids namely; Arginine, citrulline, ornithine, lysine and hydroxylysine metabolize in our body. Loss of body protein represents a typical feature of the catabolic response to surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery
* ASA II,III

Exclusion Criteria:

* Emergency surgery
* Associated renal or liver disease
* Chronic disease as D.M

Ages: 55 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiopulmonary bypass and thoracotomy for lung resection secondary to lung carcinoma, three samples will be taken to evaluate the levels of basic amino acids and NO levels
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-02 (Estimated)

PRIMARY OUTCOMES:
basic aminoacids and NO levels | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt